CLINICAL TRIAL: NCT06931093
Title: The Effectiveness of Group Guided Written Exposure Therapy for CPTSD Symptoms Among Adolescents : A Multi-centered Randomized Controlled Trail
Brief Title: The Effectiveness of Group Guided Written Exposure Therapy for CPTSD Symptoms Among Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yinyin Zang, PhD, Research Fellow, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GWE-C on Adolescents CPTSD
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: CPTSD, Compelx Post-traumatic Stress Disorder
Keywords: adolescents; randomized controlled trial; Complex PTSD

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomization will be conducted by an independent research assistant, and the random sequence will be concealed from the investigators until the process is completed. Outcome assessors will be blinded to participants' treatment conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GWE-C (Experimental)
  Interventions: Behavioral: Group Guided Written Exposure Therapy for CPTSD (GWE-C)
- Supportive counselling treatment group (ST) (Active Comparator)
  Interventions: Behavioral: Supportive counselling

INTERVENTIONS:
Behavioral: Group Guided Written Exposure Therapy for CPTSD (GWE-C) — Group Guided Written Exposure Therapy for CPTSD (GWE-C) is a manualized, exposure-based therapeutic program consisting of 7 to 10 sequential sessions. The intervention follows a structured sequence of trauma processing that addresses trauma details, associated emotions, cognitions, and impacts. Writing tasks incorporate imagery dialogues, self-compassion exercises, and resource identification to help participants alleviate C-PTSD symptoms.
  The interval between two consecutive sessions ranges from 0 to 2 days, with participants expected to complete all sessions within 1 to 2 weeks. The first and last sessions are scheduled to last 1.5 hours each, while the intermediate sessions are 60 minutes in duration. Each group will consist of 6 to 10 participants and will be facilitated by one counselor and one assistant.
  Arms: GWE-C
Behavioral: Supportive counselling — Supportive counselling, the comparator intervention, is a non-trauma-focused treatment based on the Rogerian psychotherapy model and has been used as an active comparator in previous trials of trauma-focused therapies. The program comprises seven sessions: the first two employ group activities such as card games and interactive drawing to build a sense of belonging; sessions three to six focus on stress management and emotion regulation skills through methods including expressive drawing, relaxation training, and resource identification; the final session emphasizes reflection and sharing. Throughout, counsellors provide supportive guidance to encourage emotional expression, mutual listening, and peer support, while discussions deliberately exclude participants' individual traumatic experiences.
  Arms: Supportive counselling treatment group (ST)

SUMMARY:
This study aims to examine the effectiveness of group-delivered Guided Written Exposure Therapy for Complex Post-Traumatic Stress Disorder (GWE-C) among Chinese adolescents through a randomized controlled trial. A total of 120 participants will be recruited, with 60 randomized to the GWE-C group and 60 randomized to the supportive therapy (ST) group. The GWE-C intervention will consist of 7 to 10 group sessions. The primary outcome, assessed by the International Trauma Questionnaire (ITQ), will be measured at baseline, post-treatment, 1-month follow-up, and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 10 and 18 years;
* Meet the diagnostic or subclinical criteria for Complex PTSD (C-PTSD), defined as the presence of at least one positive symptom in each of the PTSD symptom clusters, along with at least one positive symptom in each of the Disturbance in Self-Organization (DSO) symptom clusters;
* Possess sufficient literacy and language skills to complete writing-based tasks;
* Be able to understand the study procedures and complete the required assessments;
* Provide written informed consent, with consent also obtained from their legal guardians.

Exclusion Criteria:

* Presence of a severe psychiatric disorder or neurodevelopmental disorder, such as schizophrenia, bipolar I disorder, autism spectrum disorder, intellectual disability, or other severe psychiatric conditions that would interfere with study participation;
* Presence of a severe physical illness that would impair the ability to engage in the intervention;
* Suicidal ideation within the past six months;
* Ongoing exposure to traumatic events;
* Currently receiving other trauma-focused psychological treatments.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
CPTSD Symptom Severity (self-report) | baseline, post treatment(2 weeks), 6 weeks, 14 weeks
  International Trauma Questionnaire-Child and Adolescent Version (ITQ-CA; Cloitre et al.,2018 ) is a self-report measure that assesses ICD-11 PTSD and CPTSD. The measure includes 6 core items of PTSD symptom clusters (ie. re-experiencing, avoidance, sense of threat), 6 core items of Disturbances in Self-Organization (DSO) clusters (ie affective dysregulation, negative self-concept, disturbed relationships). Each item is rated from 0(not at all) to 4(extremely). The Chinese version has been demonstrated good psychometric properties (Ho et al., 2022).
CPTSD Symptom Severity(interview) | baseline, post treatment(2 weeks), 6 weeks, 14weeks
  The Child CPTSD Symptom Interview (CCSI) is a 12-item semi-structured interview developed by adapting items from the Child PTSD Symptom Scale-Interview Version for DSM-5 (CPSS-5-I) and the International Trauma Interview (ITI).The PTSD section of the CCSI includes two items for each of the three PTSD symptom clusters, following the structure of the CPSS-5-I: re-experiencing (Re), characterized by flashbacks or nightmares; avoidance (Av), referring to avoidance of internal or external reminders of the traumatic event; and a sense of current threat (Th), expressed through hypervigilance or exaggerated startle reactions.The second part assesses Disturbances in Self-Organization (DSO) symptoms, based on the structure of the ITI (Roberts et al., 2019), with two items per DSO symptom cluster.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided